CLINICAL TRIAL: NCT07115329
Title: Phase 2, Multicenter, Randomized, Double-Blind Evaluation of the Efficacy and Safety of Oral GATE-251 or Placebo for the Reduction of Symptoms of Major Depressive Disorder
Brief Title: GATE-251 or Placebo for the Reduction of Symptoms of Major Depressive Disorder With Comorbid Anxiety and Insomnia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GATE-251-C-203
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: zelquisitinel; GATE-251; N-Methyl-D-aspartate receptor positive allosteric modulator; NMDA receptor positive allosteric modulator
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Phase 2 multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed dose clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and site staff, and outcomes assessors will be blinded to treatment with GATE-251 or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GATE-251 (zelquisitinel) (Experimental): GATE-251 (zelquistinel) will be administered as a single 6 mg oral tablet one time each week for 6 weeks.
  Interventions: Drug: Zelquistinel
- Placebo (Placebo Comparator): Placebo tablet identical in appearance to the experimental treatment tablet, administered as as a single oral tablet one time each week for 6 weeks.
  Interventions: Drug: Zelquistinel

INTERVENTIONS:
Drug: Zelquistinel — Zelquistinel is a positive allosteric modulator of the N-Methyl-D-Aspartate (NMDA) receptor
  Other Names: GATE-251

SUMMARY:
The goal of this clinical trial is to learn if GATE-251 works to treat depression in adults. It will also learn about the safety of GATE-251. The main questions it aims to answer are:

Does GATE-251 reduce depression scores in participants compared to participants who take a placebo (a look-alike tablet that contains no GATE-251)?

What medical problems are observed in participants who take GATE-251?

Participants will take one tablet of GATE-251 or placebo every week for 6 weeks. Participants will visit the clinic every week of the 6 week period to have the severity of their depression evaluated.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed dose clinical trial designed to evaluate the safety and efficacy of GATE-251 versus placebo in subjects with symptoms of major depressive disorder. Each subject will participate in this study up to 98 days: up to 28 days for screening, 42 days for double-blind treatment, and a 4-week follow-up period. Subjects will return to the clinic one time each week to have the severity of their depression assessed using the Hamilton depression rating scale-17. Adverse events that occurred since the last study visit will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject.
* Aged 18 to 64 years, inclusive.
* Subject has a first episode or recurrent episode diagnosis of MDD, defined by the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), ≥3 weeks and ≤18 months. The diagnosis of MDD will be made by a central rater using the Structured Clinical Interview for DSM-5 Clinical Trials version (SCID-5-CT).
* Subject has a HDRS-17 total score of ≥18 at the Screening Visit (V1) and Baseline Visit (V2) as assessed by a central rater, with no more than a 25% change from the Screening Visit (V1) to the Baseline Visit (V2)
* Subject has HARS total score ≥15 at the Screening Visit (V1) and predose at the Baseline Visit (V2), AND
* Subject has ISI total score ≥10 at the Screening Visit (V1) and predose at the Baseline Visit (V2).
* Female subjects must meet 1 of the following:

  * Surgically sterile or at least 2 years menopausal (ie, postmenopausal is defined as a woman with the absence of menses for at least 12 consecutive months). Menopausal status is to be confirmed by assessing the follicle stimulating hormone level at Screening Visit (V1), or,
  * If a woman of childbearing potential, subject must use an acceptable method of birth control from date of Screening to the last evaluation at Day 71. Must have a documented negative point of care urine pregnancy test within 24 hours prior to first dosing.
* Male subjects, including those who are surgically sterile, must use a medically acceptable form of contraception from the time of randomization until the End of Week 6 Visit. Male subjects are strongly advised to inform female partners of the need for them to use highly effective birth control during this time period.
* Ability to understand the nature and requirements of the study and is willing to comply with the study restrictions and agree to return for the required assessments.
* Provides written informed consent to participate in the study.
* Is able to communicate with investigational site personnel, able to complete patient-reported outcome measures and in the opinion of the Investigator, can be reliably rated on assessment scales.
* Have an appropriate severity of illness of at least moderately ill corresponding to a CGI-S score of ≥4 at the Screening and Baseline Visits (V1 and V2, respectively), as assessed by a central rater.

Exclusion Criteria:

* A subject who meets any of the following criteria will be excluded from study participation:
* Evidence of treatment-resistant MDD, defined by having an inadequate response (≤25%) to 2 or more different medications approved for the treatment of MDD at an adequate dose (per locally approved label) for an adequate duration during the current episode using the Massachusetts General Hospital Antidepressant Treatment Rating Questionnaire (MGH ATRQ) assessed by a site rater.
* Current DSM-5 diagnosis of bipolar (or related disorders), antisocial personality disorder, obsessive compulsive disorder, borderline personality disorder,attention-deficit/ hyperactivity disorder, post-traumatic stress disorder, or panic attacks. Subjects not meeting full DSM-5 criteria for borderline personality disorder but exhibiting recurrent suicidal gestures, threats, or self-mutilating behaviors should also be excluded.
* Subject has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychotic features.
* Subject has a score of >4 on the CADSS at the Screening Visit (V1).
* Active seizure disorder.
* Traumatic brain injury with current signs or symptoms.
* Treatment with esketamine or ketamine, any psychedelic agent, or any experimental agent being evaluated to treat depression, whether as an antidepressant or for other use, within the past 12 months.

  o Treatment with any other experimental agents not used to treat depression within the past 3 months.
* Concomitant treatment with other Food and Drug Administration (FDA)-approved antidepressants or adjuvant agents or enhancers such as dextromethorphan, antipsychotics, mood stabilizers, sedatives, stimulants, or benzodiazepines. Subject must discontinue concomitant treatment at least 14 days prior to the Baseline Visit.

  o Subjects may continue anxiolytic agents, except for drugs that are also used to treat depression. Subjects may continue sleep aids, so long as they have been on a stable dose for at least 3 months and do not intend to change dose during the Double-Blind Treatment Period (Week 1 [Day 1] through End of Week 6). However, trazodone must be discontinued for at least 14 days prior to the Baseline Visit.
* Use of cannabis or cannabis-derived molecules, including tetrahydrocannabinol (THC), whether natural or chemically-synthesized, including hemp seed oil and cannabidiol (CBD) products (eg, gummies). Subject must discontinue the use of such products at least 14 days prior to the Baseline Visit, and THC must be below the limit of detection at the Baseline Visit.
* Positive test for any drug of abuse.
* Treated with any medical device or digital therapeutics for MDD, anxiety, insomnia, or other CNS indications within 90 days of screening in this study.
* History of electroconvulsive therapy, vagus nerve stimulation, deep brain stimulation, or repetitive transcranial magnetic stimulation within the past 5 years or has had a failure of response to electroconvulsive therapy at any time.
* Subject has clinically significant renal dysfunction as assessed by the estimated glomerular filtration rate (eGFR) <70 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration-creatinine (CKD-EPI creatinine) methodology.
* Subject has liver protein and enzyme (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, total bilirubin, lactate dehydrogenase) test result >1.5 × upper limit of normal (subjects with a diagnosis of Gilbert's Syndrome may be eligible if no liver function or enzyme test results other than total bilirubin are >1.5 × upper limit of normal).
* Subject has resting radial pulse rate (supine) <60 or >100 bpm at the Screening Visit or predose Baseline, based on a single assessment.
* Subject has resting diastolic blood pressure <50 mmHg at the Screening Visit or predose Baseline.
* Subject has PR interval >250 msec at the Screening Visit or predose Baseline, or QT corrected for heart rate by Fridericia's formula (QTcF) or QT corrected for heart rate by Bazett's formula (QTcB) interval >450 msec in males or >470 msec in females, or QRS interval >120 msec, based on a single reading.
* Evidence of alcohol abuse (>4 units of alcohol on most days; 1 unit=½ pint of beer, 1 glass of wine, or 1 ounce of hard liquor/spirits) or a positive saliva alcohol screen at Screening and predose at the Baseline Visit. Alcohol consumption should be avoided for at least 24 hours prior to Baseline Visit.
* Abuse of illicit substances by DSM-5 definition of substance use disorder within the 12 months prior to the Screening Visit.
* Use of nicotine containing products (eg, cigarettes, cigars, vaping, and pipes). Nicotine containing products must be discontinued for at least 14 days prior to randomization, and nicotine or cotinine (metabolite) must be negative at Baseline.
* Use of barbiturates. Prescribed barbiturates may be continued so long as the subject has been on a stable dose for at least 3 months and the dose may not change during the Double-Blind Treatment Period.
* HIV infection, COVID-19 infection,or active hepatitis B or C, syphilis, or other ongoing infectious disease at the Screening Visit (V1).
* Has laboratory evidence of hypothyroidism at Screening Visit (V1) as measured by thyroid stimulating hormone (TSH) and reflex free thyroxine (T4). If TSH is abnormal and reflex T4 is normal, the subject may be included.
* Has current unstable diabetes or glycosylated hemoglobin (HbA1c) >7% at Screening Visit (V1).
* Currently pregnant, planning to become pregnant during the course of the study, or nursing.
* Currently working a night shift or may be required to work night shift during the course of this study, from Screening through the End of Week 6 Visit or completion of the final polysomnography for subjects who elect to participate in the polysomnography sessions.
* Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Subject has received new onset psychotherapy or had a change in the intensity of psychotherapy within 4-weeks prior to the Screening Visit (V1).
* Currently taking prohibited prescription or over-the-counter medications including herbal therapies (eg, echinacea, ginseng, ginkgo, elderberry, turmeric, ginger, valerian, chamomile, or St John's wort) and THC- or cannabis-containing products (see Exclusion Criterion 9), which may interfere with the required study psychiatric assessments.
* History of allergy, sensitivity, or intolerance to GATE-251 or NMDAR ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
* Previously participated in this study or Study GATE-251-C-202 or currently enrolled in any other clinical study.
* Body mass index of >40 kg/m2 at the Screening Visit (V1).
* Subject is an employee of Worldwide or the Investigator or study site with direct involvement in the study or other studies under the direction of that Investigator or study site; a family member of an employee of the Investigator; or an employee of Gate Neurosciences, Inc. or a family member of an employee.
* In the opinion of the Investigator, the subject has a significant risk for suicidal behavior during the course of participation in the study, OR

  * At the Screening Visit (V1), the subject scores "Yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS with reference to a 6-month period prior to Screening Visit (V1), or
  * At the Screening Visit (V1), the subject has had 1 or more suicidal attempts with reference to a 2-year period prior to Screening Visit (V1), or
  * The subject is considered to be an imminent danger to themself or others, or
  * At the Baseline Visit (V2), the subject scores "Yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS
* The subject is judged by the Investigator or the Worldwide and Sponsor medical monitors to be appropriate for the study for any reason

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 164 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Rating Scale-17 (HDRS-17) score compared to Placebo | Change in score from baseline to 6 wweeks
  HDRS-17 is used to assess the severity of depression. The range of scores for the HDRS-17 is 0 - 52 with lower scores indicating a better outcome

SECONDARY OUTCOMES:
Change in the Clinical Global Impressions - Severity (CGI-S) score compared to placebo | Change in score from baseline to 6 weeks
  The CGI-S is a 7-level rating scale used by a clinician to gauge depression severity. The range of scores is 0-7 with lower scores indicating a better outcome

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - NoesisPharma, LLC, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Catalina Research Institute, LLC, Montclair, California
  - Excell Research, Inc, Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - Studyops Inc, San Francisco, California
  - Lumos Clinical Research Center, San Jose, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Premier Clinical Research Institute Inc, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - EquiPath Health and Research Tampa Bay, LLC, Riverview, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Denali Health Atlanta, LLC, Stone Mountain, Georgia
  - Sunstone Therapies, Rockville, Maryland
  - Continental Clinical Solutions, Towson, Maryland
  - Vitalix Clinical, Worcester, Massachusetts
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - IMA Clinical Research - NYC Midtown, New York, New York
  - IMA Clinical Research - NYC Uptown, New York, New York
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Scranton Medical Institute, LLC, Moosic, Pennsylvania
  - Adams Clinical, Philadelphia, Pennsylvania
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Synapsis Bio, Atascocita, Texas
  - Adams Clinical Dallas, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No